CLINICAL TRIAL: NCT00730041
Title: Randomized Placebo-Controlled Study of the Pillar® Palatal Implant System With CPAP
Brief Title: Palatal Implants in Combination With Continuous Positive Airway Pressure to Treat Obstructive Sleep Apnea
Acronym: Pillar-CPAP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Medtronic acquisition of Restore Medical, business decision
Sponsor: Medtronic Xomed, Inc. (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: David Hodge, Medtronic Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 845
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Results first posted 2009-11-09 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: obstructive sleep apnea; continuous positive air pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palatal Implants (Active Comparator): Pillar(R) Palatal Implants in combination with continuous positive airway pressure (CPAP) in subjects diagnosed with obstructive sleep apnea (OSA)
  Interventions: Device: Pillar Palatal Implant System
- Sham procedure (Sham Comparator): Sham (procedure but no implants inserted) in combination with continuous positive airway pressure (CPAP) in subjects diagnosed with obstructive sleep apnea (OSA)
  Interventions: Device: Sham system

INTERVENTIONS:
Device: Pillar Palatal Implant System — The Pillar system is intended as an initial treatment option for mild to moderate OSA. It consists of a delivery system and an implant. The delivery system is comprised of a disposable handle and needle assembly that allows for positioning and placement of the implant within the soft palate of the mouth. The 18mm x 2mm implant is a cylindrical shaped segment of braided polyester filaments that is intended for permanent implantation into the soft palate. The implant is pre-loaded into the needle. Three implants are placed in each subject under local anesthesia. Because implants are not able to be seen in the soft palate tissue, the physician is unable to see if an implant is placed or not placed and thus is blinded to the intervention type.
  Other Names: soft palate implants; palatal implants
  Arms: Palatal Implants
Device: Sham system — The Pillar system consists of a delivery system and an implant. The only difference between the treatment and sham arm in this study is that the sham delivery device is not pre-loaded with the implant. Otherwise the appearance, manufacturing and function of the delivery devices are identical. Three insertions are made, but no implants are actually deployed during the procedure. Because implants are not able to be seen in the soft palate tissue, the physician is unable to see if an implant is placed or not placed and thus is blinded to the intervention type.
  Other Names: soft palate implants; palatal implants
  Arms: Sham procedure

SUMMARY:
The study will be done for the following purposes:

* to see if Pillar implants in combination with CPAP therapy can help people with their OSA by decreasing the CPAP pressures
* to find out if receiving Pillar implants will increase CPAP use

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is the intermittent cessation of breathing during sleep due to the collapse of the pharyngeal airway. As reported in the April 2004 Journal of the American Medical Association, it is estimated that 59 million people in the United States suffer OSA symptoms. OSA is typically diagnosed through an overnight sleep study (polysomnogram or PSG) in a sleep laboratory or a portable monitoring system. The American Academy of Sleep Medicine's (AASM) recommended treatment for patients with OSA is Continuous Positive Airway Pressure (CPAP), which is a life-long therapy that requires subjects to wear a nasal or facial mask connected to a portable airflow generator while sleeping. CPAP therapy is intended to treat OSA by preventing collapse of the upper airway during sleep with the use of positive pressure. Compliance with CPAP therapy may be a problem as fewer than 50% of patients using CPAP have been considered "regular" users due to a variety of factors such as claustrophobia, nasal stuffiness, social factors, and inconvenience.

The Pillar® Palatal Implant System is currently commercially available in the United States, Europe, and other countries to treat habitual snoring and mild to moderate OSA. It is a minimally invasive, well-tolerated procedure that reduces the flexibility of the soft palate and increases its stiffness, which reduces snoring and may limit the palate's ability to collapse into the airway during sleep contributing to clinical episodes of OSA.

The Pillar system consists of a delivery system and an implant. The delivery system is comprised of a disposable handle and needle assembly that allows for positioning and placement of the implants within the soft palate. The 18mm x 2mm implant is a cylindrical shaped segment of braided polyester filaments that is intended for permanent implantation into the soft palate. The needle of the delivery system is inserted into the soft palate, near the hard palate junction. A sliding thumb switch is retracted to deploy the implant. The first implant is placed midline and two additional implants are placed, one on each side approximately 2mm from the midline implant, for a total of three implants.

An antiseptic rinse is recommended pre-procedure and an appropriate broad-spectrum antibiotic should be given both pre and post-procedurally. Local anesthesia is used in all patients. Pain medication is suggested to manage discomfort in the immediate post-operative period.

While the Pillar procedure can be effective in the treatment of mild to moderate OSA, its effect in combination with CPAP treatment has never been studied. In this study, the treatment of OSA using the Pillar procedure in combination with standard CPAP treatment vs. sham procedure in combination with standard CPAP treatment will be investigated. All subjects will be asked to continue their normal use of CPAP treatment during the study. The study will evaluate whether or not the Pillar implants allow less therapeutic pressure to be used in treating the OSA and if less pressure translates to increased usage.

ELIGIBILITY:
Inclusion Criteria:

* OSA documented by sleep study demonstrating AHI > 10, where hypopneas are defined by Medicare criteria requiring a 4% desaturation
* Adequate CPAP therapy titration (residual AHI < 5) resulting in a therapeutic pressure ≥7 cm H20 from baseline PSG
* Currently using or willing to change to Respironics CPAP device (without A-flex, C-flex and Bi-flex enabled) with SmartCard technology
* Currently dissatisfied with CPAP therapy

Exclusion Criteria:

* Uses full face mask
* Soft palate length insufficient to accommodate 18mm implants as measured from the hard palate junction to the base of the uvula (<25 mm)
* Drug abuse or alcoholism in the year prior to enrollment as assessed by history
* Inconsistent use of sleeping medications (1 or 2 nights per week)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Rapoport, MD, Principal Investigator — NYU Sleep Disorders Center
Locations (7):
- United States (7):
  - Arkansas Center for Sleep Medicine, Little Rock, Arkansas
  - Alta Bates Summit Medical Center, Berkeley, California
  - Sleep Center at National Jewish Medical Center, Denver, Colorado
  - Louisiana Sleep Foundation, Baton Rouge, Louisiana
  - Regions Hospital; Health Partners Sleep Health Center, Saint Paul, Minnesota
  - NYU Sleep Disorders Center, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All initial study candidates were recruited from the Investigator's general patient population and related physician referral base. The Investigator or designee screened each candidate to ensure that all inclusion and exclusion criteria were met.
Pre-assignment Details: After initial screening, all subjects had a polysomnogram (PSG) with continuous positive airway pressure (CPAP) titration to determine the therapeutic pressure. Subjects collected a minimum of two weeks of SmartCard data using CPAP machine prior to the intervention in order to establish baseline usage info. Group was determined at the intervention.
Groups:
- Pillar(R) Palatal Implants: Pillar Implants in combination with continuous positive airway pressure (CPAP)
- Sham Procedure With no Implants: Sham (procedure but no implants inserted) in combination with continuous positive airway pressure (CPAP)
Period: Overall Study
Arm/Group | Pillar(R) Palatal Implants | Sham Procedure With no Implants
Started | 26 (4/26 (15.4%) female, 22/26 (84.6%) male) | 25 (4/25 (16.0%) female, 21/25 (84.0%) male)
Completed | 26 | 23 (One subject did not return for the final PSG or final visit, and one missed only the final visit.)
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pillar(R) Palatal Implants | Sham Procedure With no Implants | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 3 | 2 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 52.3 (10.3) | 51.1 (9.0) | 51.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 22 | 21 | 43
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Pressure From a Polysomnogram (PSG) With Continuous Positive Airway Pressure (CPAP) Titration
Description: The American Academy of Sleep Medicine's (AASM) recommended treatment for patients with obstructive sleep apnea (OSA) is Continuous Positive Airway Pressure (CPAP), which is a life-long therapy that requires subjects to wear a nasal or facial mask connected to a portable airflow generator while sleeping. CPAP therapy is intended to prevent collapse of the upper airway. CPAP pressures are measured in centimeters of water, and range in whole numbers from 4cm H2O to 20cm H2O. The therapeutic pressure is usually determined during overnight polysomnography and usually performed by a technician.
Time Frame: Baseline and 3 months post-procedure
Population: 50 of 51 total participants returned to the sleep lab for the 90-day PSG. All 50 participants are part of the primary endpoint analysis.
Measure: Mean (Standard Deviation); unit: centimeters of water (cm H2O)
Arm/Group | Pillar(R) Palatal Implants | Sham Procedure With no Implants
Number analyzed (Participants) | 26 | 24
centimeters of water (cm H2O)
  Assigned Pressure at Baseline | 10.9 (2.7) | 10.9 (2.6)
  Assigned Pressure at 90 days | 10.3 (2.4) | 9.8 (3.0)

2. Secondary Outcome: Visual Analog Scale (VAS) for Continuous Positive Airway Pressure (CPAP) Comfort Score.
Description: The candidate was asked to complete a questionnaire that included a VAS describing CPAP therapy comfort. Scores ranged from 0 (very uncomfortable) to 10 (very comfortable).
Time Frame: Baseline and 4 months post-procedure
Population: Two participants in the sham group became lost to follow-up and did not return for the final follow-up.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Pillar(R) Palatal Implants | Sham Procedure With no Implants
Number analyzed (Participants) | 26 | 23
Scores on a Scale
  Baseline Score | 3.5 (2.1) | 3.2 (1.8)
  Post 90-day PSG Score (4 months post-procedure) | 5.6 (2.5) | 4.3 (3.2)

3. Secondary Outcome: Measurement of Total Leak as Recorded by SmartCard (Home Compliance Feature of the Continuous Positive Airway Pressure Machine)
Description: Leak is an indicator of mask/headgear fit and can also be used to substantiate or contradict an assigned therapeutic pressure. Total leak is the sum of intentional leak to prevent carbon dioxide rebreathing and unintentional leak. Each mask has a known amount of leak (the intentional leak), and subjects were instructed not to changes masks to minimize this variable. Approximate range is 0-100, and the amount of leak increases as the number increases. Average leak values are in the 20-50 liters per minute range. The CPAP machine records leak data during each night of usage and can average.
Time Frame: Baseline and 4 months post-procedure
Population: Five participants in the sham group did not return their SmartCards at the final study visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pillar(R) Palatal Implants | Sham Procedure With no Implants
Number analyzed (Participants) | 26 | 20
Units on a scale
  Baseline Score | 46.8 (15.1) | 47.2 (7.2)
  Post 90-day PSG Score (4 months post-procedure) | 48.8 (18.4) | 50.8 (10.6)

4. Secondary Outcome: Visual Analog Scale (VAS) to Measure Continuous Positive Airway Pressure (CPAP) Satisfaction.
Description: The candidate was asked to complete a questionnaire that included a VAS describing CPAP satisfaction. Scores ranged from 0 (very unsatisfied) to 10 (very satisfied).
Time Frame: Baseline and 4 months post-procedure
Population: Two participants in the sham group became lost to follow-up and did not return for the final follow-up.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Pillar(R) Palatal Implants | Sham Procedure With no Implants
Number analyzed (Participants) | 26 | 23
Scores on a Scale
  Baseline Score | 3.8 (2.3) | 4.2 (2.2)
  Post 90-day PSG Score (4 months post-procedure) | 6.5 (2.3) | 5.0 (3.1)

5. Secondary Outcome: Epworth Sleepiness Scale (ESS), a Validated Measure of Daytime Sleepiness.
Description: The Epworth Sleepiness Scale (ESS) was included in the subject questionnaire as a tool to further assess the quality of sleep for each subject throughout the follow-up period. This scale is a validated clinical indicator that quantifies the patient's chance of falling asleep during eight different activities of daily living such as reading, talking, resting and driving. Each of the eight questions has four possible responses: 0 = would never doze, 1 = slight chance of dozing, 2 = moderate chance of dozing to 3 = high chance of dozing, for a possible maximum score of 24.
Time Frame: Baseline and 4 months post-procedure
Population: Two participants became lost to follow-up and did not return for the final study visit.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Pillar(R) Palatal Implants | Sham Procedure With no Implants
Number analyzed (Participants) | 26 | 23
Scores on a Scale
  Baseline Score | 10.7 (5.7) | 11.3 (5.9)
  Post 90-day PSG Score (4 months post-procedure) | 7.9 (5.2) | 9.7 (4.8)

6. Secondary Outcome: Functional Outcomes of Sleep Questionnaire (FOSQ), a Validated Measure the Impact of Excessive Sleepiness on Multiple Activities of Daily Living.
Description: The FOSQ can assess the quality of sleep and this scale is a validated measure the impact of excessive sleepiness on multiple activities of daily living. It has 30 questions in 5 subgroups of general productivity (8 questions), social outcome (2), activity level (9), vigilance (7), and intimate relationships and sexual activity (4). Responses for each question range from 1 (extreme difficulty or low activity level) to 4 (no difficulty or high activity level) for each subgroup. A mean is calculated for each subgroup, and then the mean of the subgroups is calculated and multiplied by 5.
Time Frame: Baseline and 4 months post-procedure
Population: Two subjects became lost to follow-up and did not return for the final study visit.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Pillar(R) Palatal Implants | Sham Procedure With no Implants
Number analyzed (Participants) | 26 | 23
Scores on a Scale
  Baseline Score | 15.5 (2.9) | 15.5 (3.1)
  Post 90-day PSG Score (4 months post-procedure) | 17.4 (2.4) | 16.0 (3.1)

7. Secondary Outcome: Measurement of Usage (Hours) of the Continuous Positive Airway Pressure Machine as Recorded by SmartCard (Home Compliance Monitor)
Description: The CPAP machine has an internal clock/calendar, and capabilities to record usage onto a removable data card the size of a credit card. Data is recorded from the first time the machine is turned on to the last time the machine is turned on during a given period in which the SmartCard is present in the machine. The SmartCard records all days during the given period and keeps track of days in which the CPAP machine is used and days in which it is not used. The SmartCard data is able to be downloaded to a computer for review and analysis.
Time Frame: Baseline and 4 months post-procedure
Population: Five participants in the sham group did not return their SmartCards at the final study visit.
Measure: Mean (Standard Deviation); unit: Average hours per day of days used
Arm/Group | Pillar(R) Palatal Implants | Sham Procedure With no Implants
Number analyzed (Participants) | 26 | 20
Average hours per day of days used
  Baseline Usage | 6.0 (2.5) | 5.2 (1.9)
  Post 90-day PSG Usage (4 months post-procedure) | 6.0 (2.4) | 5.2 (2.1)

ADVERSE EVENTS:
Time Frame: 4 months (from implant to the subject's final follow-up visit at approximately 4 months post-implant procedure)
Description: Subjects were asked at the 7 day follow-up and the 4 month follow-up about any changes in health they experienced since the implant/sham procedure. They were also instructed to contact the study physician or coordinator if they had any problems between visits. Each subject's medical records were reviewed for adverse events at monitoring visits.
Arm/Group | Pillar(R) Palatal Implants | Sham Procedure With no Implants
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 17/26 | 9/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pillar(R) Palatal Implants (N=26) | Sham Procedure With no Implants (N=25)
Sore or scratchy throat at site of needle insertion (Injury, poisoning and procedural complications) | 13 (13) | 7 (7) — Note that these reported adverse events occurred shortly after the procedure and were not associated with cold or flu symptoms. All resolved on their own or with the short-term use of pain medication.
Mild bleeding at the site of needle insertion during the procedure (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) — All occurrences resolved the same day with minimal or no intervention by the study physician.
Medication reaction (non-study related, non-life threatening) (General disorders) | 2 (2) | 1 (1) — These reactions were caused by medications the subjects took outside of the study related treatment and resulted in 2 cases of hives and 1 headache with hypertension and lasted briefly.
Sinus infection (Infections and infestations) | 2 (2) | 0 (0) — Not related to the subject's participation in this study.

LIMITATIONS AND CAVEATS:
The study was underpowered for this comparison as only half the planned enrollment occurred. Also, changes occurred with the sleep stage and position as well as the masks used between the two PSGs, which may have affected some of the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agree to submit copies of proposed manuscripts or abstracts to sponsor at least 45 days in advance of public release. If sponsor requests or requires changes, an additional 90 days are allowed for this. Upon completion of the last subject follow-up for the Evaluation, a period of one year shall be reserved for publication of the entire trial results. No individual investigator may publish their individual site results prior to the publication of the group data.